CLINICAL TRIAL: NCT06921187
Title: Etude de la Perception Auditive après Exposition PROgressive Aux Sons Aversifs Chez Des Personnes MISophonEs
Brief Title: Study of Auditory Perception After Progressive Exposure to Aversive Sounds in People With Misophonia
Acronym: PROMISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-058; 2024-A02048-39 (Other: ID-RCB)
Record Dates: First submitted 2025-03-18; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Misophonia
MeSH Terms: conditions — misophonia

STUDY DESIGN:
Intervention Model Description: exposure to unpleasant sounds at home is the focus of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Behavioral: Psychoacoustic test; Other: semi-structured interviews
- Misophonia group (Experimental)
  Interventions: Behavioral: Psychoacoustic test; Other: semi-structured interviews; Other: Exposure to unpleasant sounds

INTERVENTIONS:
Behavioral: Psychoacoustic test — Natural sounds will be presented at different decibels (dB), and the subject will be asked to rate the pleasantness/unpleasantness of the sound heard on a visual analogue scale, as well as the loudness (subjective intensity) of the sound heard.
Other: semi-structured interviews — interview, designed under the supervision of a psychologist and using the methodology of micro-phenomenological interviews the aim of these interviews is to gain access to the participants' experiences, as they describe them in the first person, during misophonic episodes
Other: Exposure to unpleasant sounds — Home exposure is a practice whereby participants voluntarily subject themselves to SMs in a controlled environment.
  Participants will be asked to complete two tasks: firstly, they will have to expose themselves to all 10 sounds at least twice a week; secondly, they will have to record the annoyance felt for each sound and the subjective loudness (loudness) of each SM using VAS.
  Arms: Misophonia group

SUMMARY:
The primary objective of the project is to characterise and measure the auditory perception of subjects with misophonia compared with the auditory perception of control subjects.

ELIGIBILITY:
Inclusion Criteria:

For all participants

* Obtain oral consent from the participant after receiving information about the study,
* Be 18 years or older on the day of inclusion,
* Be fluent in French (spoken and written),
* Have no known hearing loss, verified by pure tone audiometry.
* Declare that they do not have tinnitus,
* Declare that they do not have hyperacusis, verified by measuring discomfort thresholds.
* Be affiliated to the social security or equivalent scheme.

For participants with misophonia:

- Declare discomfort, reduced tolerance to specific sounds (mouth noises, throat clearing, breathing, etc.).

Exclusion Criteria:

* Bear the after-effects of an ear infection and/or have a history of an ENT disease that permanently affects hearing or balance (vestibular schwannoma, Ménière's disease, sudden or fluctuating deafness, congenital hypoacusis),
* Be under guardianship,
* deprived of liberty by judicial or administrative decision, or subject to legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
score on a visual analogue scale from 0 (pleasant sound) to 10 (unpleasant sound) | 1 week after enrollment
  sounds will be presented at different decibels and the subject will be asked to rate the pleasantness/unpleasantness of the sound on a visual analogue scale
score on a visual analogue scale from 0 (very low intensity) to 10 (extremely intense) | 1 week after enrollment
  sounds will be presented at different decibels and the subject will be asked to rate the intensity of the sound on a visual analogue scale

SECONDARY OUTCOMES:
Measuring the consistency of the psychoacoustic test | 1 week after enrollement
  consistency measured by calculating Cronbach's alpha coefficient
the number of redundant themes in the semi-structured interviews | 1 month after enrollment
  the interviews consist of open-ended questions covering different aspects of the experiences of misophone subjects
score on a visual analogue scale from 0 (very little discomfort) to 10 (extreme discomfort) | 1 month after enrollment and 2 months after enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de Recherche en Psychologie et Neuroscience (CRPN), Marseille
  - CEntre de Recherche et d'Innovation en Audiologie Humaine, Paris

IPD SHARING:
Plan to Share IPD: Undecided